CLINICAL TRIAL: NCT05832554
Title: Comparison of the Effects of Nasopharyngeal and Oropharyngeal Airway Use on Gastric Insufflation in Patients Who Are Expected to Have Difficult Mask Ventilation
Brief Title: Comparison of the Effects of Nasal and Oral Airway Use on Gastric Insufflation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Diskapi Teaching and Research Hospital (Other)
Responsible Party: Principal Investigator, derya özkan, Professor MD, Diskapi Teaching and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: AESH-2023-002
Record Dates: First submitted 2023-04-15; First posted 2023-04-27 (Actual); Last update posted 2024-07-25 (Actual); Status verified 2024-07

CONDITIONS: Gastric Insufflation; Difficult Mask Ventilation
Keywords: Nasopharyngeal airway; Oropharyngeal airway; Difficult airway
MeSH Terms: interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nasopharyngeal airway (Active Comparator): Patients with nasopharygeal airway placed
  Interventions: Device: nasal airway
- Orophryngeal airway (Active Comparator): Patients with oropharygeal airway placed
  Interventions: Device: oral airway

INTERVENTIONS:
Device: nasal airway — nasopharyngeal airway
  Arms: Nasopharyngeal airway
Device: oral airway — oropharyngeal airway
  Arms: Orophryngeal airway

SUMMARY:
The goal of this clinical trial is to compare the effects of nasopharyngeal and oropharyngeal airway on gastric insufflation in patients undergoing general anesthesia and expected difficult mask ventilation. The main questions it aims to answer are:

* Is there a difference between the presence of gastric insufflation in the use of nasopharyngeal and oropharyngeal airways?
* Is there a difference between the antral area sizes measured before and after ventilation After general anesthesia induction, nasopharyngeal or oropharyngeal airway will be placed in participants and real-time ultrasonographic gastric antral area imaging will be performed during mask ventilation. Researchers will compare the effects of nasopharyngeal and oropharyngeal airway use on gastric insufflation.

DETAILED DESCRIPTION:
Patients who are expected to have difficult mask ventilation and receive general anesthesia will be included in the study. After preoperative gastric antral area measurements of the patients by ultrasonography, preoxygenation will be applied and anesthesia induction will be performed. Real-time gastric ultrasonography will be performed during pressure-controlled mask ventilation for 2 minutes after nasopharyngeal or oropharyngeal airway insertion, and then antral area measurement will be repeated. After the trachea was intubated, the antral area measurement was once again performed. At the 30th, 60th, 90th and 120th seconds of ventilation, patients' SpO2, EtO2, EtCO2, peak airway pressure, tidal volume, leak volumes and hemodynamic changes will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Patients receiving general anesthesia
* ASA score I-II-III
* At least 3 criteria out of 5 difficult mask criteria defined by Langeron et al.

Exclusion Criteria:

* Patients who did not give informed consent
* Risk of aspiration
* Respiratory disease
* Facial, oropharyngeal or nasopharyngeal pathology
* Pregnancy

Ages: 18 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2023-11-24 (Actual); Study Completion 2024-01-05 (Actual)

PRIMARY OUTCOMES:
Presence of gastric insufflation | During 2 minutes mask ventilation
  Presence of gastric insufflation by ultrasound imaging in nasopharyngeal and orophrayngeal airway use
Difference in antral area sizes | During 2 minutes mask ventilation
  Difference in antral area sizes measured by ultrasound imaging before and after ventilation

SECONDARY OUTCOMES:
Leakage volume | During 2 minutes mask ventilation
  Leakage volume per minute in nasopharyngeal and orophrayngeal airway use

CONTACTS AND LOCATIONS:
Overall Officials: Derya Ozkan, proff MD, Principal Investigator — Ankara Etlik City Hospital
Locations (1):
- Ankara Etlik City Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bouvet L, Albert ML, Augris C, Boselli E, Ecochard R, Rabilloud M, Chassard D, Allaouchiche B. Real-time detection of gastric insufflation related to facemask pressure-controlled ventilation using ultrasonography of the antrum and epigastric auscultation in nonparalyzed patients: a prospective, randomized, double-blind study. Anesthesiology. 2014 Feb;120(2):326-34. doi: 10.1097/ALN.0000000000000094. PMID 24317204
- [Background] Langeron O, Masso E, Huraux C, Guggiari M, Bianchi A, Coriat P, Riou B. Prediction of difficult mask ventilation. Anesthesiology. 2000 May;92(5):1229-36. doi: 10.1097/00000542-200005000-00009. PMID 10781266